CLINICAL TRIAL: NCT00528658
Title: Cost-effectiveness Analysis of Oral Paracetamol and Ibuprofen for Treating Pain After Soft Tissue Limb Injuries: Double-blind, Randomised Controlled Trial
Brief Title: Cost-effectiveness of Two Painkillers for Treating Pain After Limb Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Academy of Medicine (Other)
Responsible Party: Principal Investigator, Colin Graham, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKCEM06-07/DG2041095; HKCEM Grant 2006-07; CUHK DG 2041095
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Soft Tissue Injuries
Keywords: Soft Tissue Injuries
MeSH Terms: conditions — Soft Tissue Injuries | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Paracetamol; Drug: Ibuprofen placebo
- 2 (Experimental)
  Interventions: Drug: Ibuprofen; Drug: Paracetamol Placebo
- 3 (Experimental)
  Interventions: Drug: Paracetamol; Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol — 1g qid
  Arms: 1; 3
Drug: Ibuprofen — 400mg tid
  Arms: 2; 3
Drug: Paracetamol Placebo — equivalent to 1g qid
  Arms: 2
Drug: Ibuprofen placebo — Equivalent to 400mg tid
  Arms: 1

SUMMARY:
Background: Paracetamol and non-steroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen are commonly used oral analgesics in emergency departments (ED) not only in Hong Kong but throughout the world. There are no large-scale (n>100), prospective, randomised studies comparing paracetamol with ibuprofen in the management of acute soft tissue injury.

As paracetamol is cheaper than most NSAIDs, may be as effective in the management of acute pain and possibly with fewer adverse effects, a large-scale, randomised, controlled trial is needed to answer questions of relative analgesic efficacy, safety and cost-effectiveness. Previous comparative studies on NSAIDS have been done in this unit and have suggested equivalence between two NSAIDs and paracetamol, but numbers were small and drug doses were modest.

Objective: To compare the efficacy, safety and cost between oral ibuprofen and paracetamol in pain control for acute soft tissue injuries in an ED setting

Design: Prospective, double-blind, randomised controlled trial with three arms: oral paracetamol with placebo; oral ibuprofen with placebo; paracetamol and ibuprofen in combination

Participants: 783 subjects having sustained isolated soft tissue limb injury without significant fracture presenting to the ED of Prince of Wales Hospital

Main outcome measures: Pain relief profiles of paracetamol, ibuprofen and the combination of both; adverse effect profiles of paracetamol, ibuprofen and the combination of both; overall cost effectiveness of paracetamol, ibuprofen and the combination of both from the perspective of the healthcare provider

ELIGIBILITY:
Inclusion Criteria:

* All patients >16 years presenting to the ED with isolated soft tissue injury without significant fracture
* between 9am to 5pm, Monday to Friday,

Exclusion Criteria:

* History of :

  * peptic ulceration or hemorrhage
  * recent anticoagulation
  * pregnancy
  * adverse reaction to paracetamol or ibuprofen
  * renal or cardiac failure
  * hepatic problems
  * rectal bleeding
  * chronic NSAID consumption
  * asthma
  * chronic obstructive pulmonary disease
  * chronic pain syndromes
  * prior treatment with analgesia for the same injury
  * physical, visual or cognitive impairment making use of the visual analogue scale unreliable

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
analgesic efficacy both at rest and with movement | 72 hours

SECONDARY OUTCOMES:
presence, frequency and duration of adverse effects; cost-effectiveness analysis; patient satisfaction with analgesia | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Graham, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong

REFERENCES:
- [Derived] Hung KKC, Graham CA, Lo RSL, Leung YK, Leung LY, Man SY, Woo WK, Cattermole GN, Rainer TH. Oral paracetamol and/or ibuprofen for treating pain after soft tissue injuries: Single centre double-blind, randomised controlled clinical trial. PLoS One. 2018 Feb 6;13(2):e0192043. doi: 10.1371/journal.pone.0192043. eCollection 2018. PMID 29408866